CLINICAL TRIAL: NCT01672138
Title: PVAI Plus Scar Homogenization and Ablation of Non-PV Triggers Ensure Long-term Recurrence-free Survival in Non-paroxysmal Atrial Fibrillation
Brief Title: Pulmonary Vein Antrum Isolation (PVAI) Plus Scar Homogenization and Non-PV Triggers Ensure Long-term Recurrence-free Survival in Non-paroxysmal Atrial Fibrillation
Acronym: TANTRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Collaborators: RCCS Monzino Hospital, Milan, Italy (Unknown); Ospedale dell'Angelo, Venezia-Mestre (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive medical director, TCAI, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TANTRA_TCAI
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Persistent Atrial Fibrillation; Long-standing Persistent Atrial Fibrillation
Keywords: PVAI; NPAF; Non-PV triggers
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): Pulmonary Vein Antrum Isolation (PVAI) + isolation of left atrial posterior wall
  Interventions: Procedure: Pulmonary Vein Antrum Isolation
- Study I (Active Comparator): PVAI+ scar homogenization
  Interventions: Procedure: Pulmonary Vein Antrum Isolation; Procedure: scar homogenization
- Study II (Active Comparator): PVAI + isolation of left atrial posterior wall + non-PV triggers ablation
  Interventions: Procedure: Pulmonary Vein Antrum Isolation; Procedure: scar homogenization; Procedure: Non-PV triggers ablation

INTERVENTIONS:
Procedure: Pulmonary Vein Antrum Isolation — Radio-frequency catheter ablation of pulmonary vein antrum extended to the left atrial posterior wall
  Other Names: PVAI
Procedure: scar homogenization — PVAI + RF energy will be delivered until all abnormal potentials in the low-voltage areas are eliminated.
  Arms: Study I; Study II
Procedure: Non-PV triggers ablation — PVAI + Isolation of LA posterior wall + Catheter ablation of triggers originating from extra-PV sites
  Arms: Study II

SUMMARY:
This study aims to examine the long-term success rate of catheter ablation in non-paroxysmal atrial fibrillation patients using different ablation strategies such as : (i) pulmonary vein antrum isolation (PVAI) + isolation of left atrial posterior wall, (ii) PVAI plus scar homogenization, (iii) PVAI plus isolation of posterior wall plus ablation of non-PV triggers [ PVAI: Pulmonary Vein Antrum Isolation

Non-PV triggers: Triggers arising from sites other than pulmonary veins]

DETAILED DESCRIPTION:
Back ground: Pulmonary vein antrum isolation (PVAI) as a lone procedure, is known to have limited success rate in terms of long-term recurrence-free survival in non-paroxysmal atrial fibrillation (NPAF) and additional ablations isolating extra-PV triggers seem to improve the outcome (1). The extra-PV triggers include triggers from other sites such as left atrial posterior wall, superior vena cava, interatrial septum, crista terminalis, left atrial appendage and coronary sinus (1, 2). These are known to be independent predictors of late AF recurrence following catheter ablation (3, 4, and 5). Earlier studies have demonstrated better ablation outcome in NPAF when non-PV triggers sites were isolated along with PVAI (5, 6). Moreover, Verma et al had reported high (57%) recurrence rate post-index procedure in AF patients with pre-existent scar (7). However, published data are conflicting regarding the benefits of additional substrate guided ablation (scar homogenization) compared to conventional PVAI alone strategy (8). Also, limited data is available showing a comparison of the lasting efficacy of the above three procedures when used in different combinations.

Hypothesis: The combined ablation strategy including PVAI, scar homogenization and ablation of extra-PV triggers has the highest likelihood of maintaining long-term sinus rhythm in patients with NPAF.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients undergoing first catheter ablation for drug-refractory Persistent (PerAF) or long-standing persistent AF (LSPAF)
3. Ability to understand and provide signed informed consent

Exclusion Criteria:

1. Previous catheter ablation or MAZE procedure in left atrium
2. Reversible causes of atrial arrhythmia such as hyperthyroidism, sarcoidosis, pulmonary embolism etc

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial arrhythmia | 3 years
  Any episode of AF/AT (atrial tachycardia) longer than 30 seconds will be considered as recurrence). Episodes that occur during the first 3 months of the procedure (blanking period) will not be considered as recurrence.

SECONDARY OUTCOMES:
Improvement in quality of life | 3 years
  Improvement in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — TCAI
Locations (2):
- United States (2):
  - St. david's medical Center, Austin, Texas
  - Texas Cardiac arrhythmia Institute, St. David's Hospital, Austin, Texas